CLINICAL TRIAL: NCT06698302
Title: Validation of COMPAT-SF Spanish Translation
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 009.GID.2024.D
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Questionnaires — Administer translated COMPAT-SF questionnaires to Spanish-speaking CP patients

SUMMARY:
Prospective translation validation pilot study that will collect data from Spanish-speaking CP patients seen at Methodist Dallas Medical Center (MDMC) beginning June 2024 through July 2027, in order to validate a Spanish-translated COMPAT-SF instrument.

DETAILED DESCRIPTION:
Prospective translation validation pilot study that will collect data from Spanish-speaking CP patients seen at Methodist Dallas Medical Center (MDMC) beginning June 2024 through July 2027, in order to validate a Spanish-translated COMPAT-SF instrument.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older in age
* Have a definite CP diagnosis and a stable pain pattern with no new interventions or medications in the last three months
* Able to read and understand the study information in Spanish
* Personally signed and dated ICF indicating that the subject has been informed of all pertinent aspects of the study
* Subject is willing and able to comply with the scheduled questionnaires

Exclusion Criteria:

* Subjects who do not meet the criteria in section 4.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spanish speaking subjects with CP diagnosis and a stable pain pattern with no new interventions or medications in the last three months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-09-13 (Estimated); Study Completion 2026-09-13 (Estimated)

PRIMARY OUTCOMES:
Face validity: | through study completion, up to 18 months
  Patient-reported feedback through a questionnaire concerning the feasibility of the translated COMPAT-SF questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Dallas Medical Center- Clinical Research Institute, Dallas, Texas, United States